CLINICAL TRIAL: NCT03543527
Title: Observational Multicenter Study of Refractory and/or Relapsing Takayasu Arteritis START: Study of Refractory and/or Relapsing TAkayasu aRTeritis
Brief Title: Study of Refractory and/or Relapsing TAkayasu aRTeritis
Acronym: START
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: START_001
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Systemic Vasculitis; Arteritis, Takayasu; Arteritis
MeSH Terms: conditions — Systemic Vasculitis; Takayasu Arteritis; Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Takayashu
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Takayasu arteritis (TA) is a vasculitis of unknown origin, resulting in progressive thickening and stenosis of large and medium arteries (the aorta and its major branches, and the pulmonary arteries). First line therapy of TA consists of high dose corticosteroids (CS) (Mukhtyar et al, 2009). Between 20 and 50% of cases respond to CS alone, with subsequent resolution of symptoms and stabilization of vascular abnormalities (Shelhamer et al, 1985; Maksimowicz-McKinnon et al, 2007). Although second-line agents (methotrexate, azathioprine, mycophenolate mofetil, cyclophosphamide) may result in initial remission, relapses remain common when prednisone is tapered (Maksimowicz-McKinnon et al, 2007). Thus, 50% of CS-resistant or relapsing TA patients may achieve sustained remission with the addition of methotrexate (Hoffman et al, 1994). During the last decade, biologics such as anti-tumor necrosis factor alpha (anti-TNFα) and anti-interleukin-6 (anti-IL-6) have been used as third-line treatment in refractory or relapsing TA. Almost 90% of CS-methotrexate resistant TA cases responded to infliximab, an anti-TNFα, and sustained remission was obtained in 37 to 76% of the cases (Schmidt et al, 2012; Comarmond et al, 2012; Mekinian et al, 2012). Tocilizumab, an anti-IL-6 has given similar results with 68% of sustained remission in refractory TA (Abisror et al, 2013). Irrespective of classical cardiovascular risk factors, the systemic inflammation and CS use play a pivotal role in the occurrence of cardiovascular thrombotic events (CVEs) (Roubille et al, 2015). As CVEs overlap with TA complications it is primordial to drastically taper CS in that vasculitis. We therefore aim to analyses prospectively the long term outcome of refractory/relapsing TA patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Takayasu arteritis according to the international criteria of the American College of Rheumatology (ACR) (Arend et al, 1990) and/or Ishikawa criteria modified by Sharma.
* Active disease according to the international criteria of the National Institute of Health (NIH) (Kerr et al, 1994)
* Able and willing to give informed consent and comply with the requirements of the study protocol

Exclusion Criteria:

* Aortitis of other cause (i.e. infectious, ANCA vasculitis, histiocytosis, cancer..)
* Lack of affiliation to a social security benefit plan (as a beneficiary or assignee)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Takayasu Patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with prednisone ≤ 0.1mg/kg per day and sustained inactive disease. | 6 months
  Proportion of patients with prednisone ≤ 0.1mg/kg per day and sustained inactive disease.

SECONDARY OUTCOMES:
incidence of relapse | 6 months
  incidence of relapse
incidence of relapse | 12 months
  incidence of relapse
incidence of treatment failure | 6 months
  incidence of treatment failure
incidence of treatment failure | 12 months
  incidence of treatment failure
incidence of revascularization procedures | 6 months
  incidence of revascularization procedures
incidence of revascularization procedures | 12 months
  incidence of revascularization procedures
incidence of adverse events of treatments received | 6 months
  incidence of adverse events of treatments received
incidence of adverse events of treatments received | 12 months
  incidence of adverse events of treatments received

CONTACTS AND LOCATIONS:
Locations (1):
- La pitié Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided